CLINICAL TRIAL: NCT01289145
Title: Stage-based Exercise Promotion Study
Acronym: STEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Responsible Party: Prof. Dr. Ralf Schwarzer, Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STEP-2011-PK
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2011-02

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
Keywords: Action Planning; Positive Outcome Expectancies; Randomized Controlled Trial; Stages of change; Health behavior; Motivation
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Participants will be allocated to a motivational intervention, a volitional intervention or the active control group.
  The motivational intervention promotes positive outcome expectancies on physical activity. The volitional intervention promotes the formulation of action plans for physical activity. Participants in the active control group, receive a quiz on physical activity and sports.
  Interventions: Behavioral: Motivational intervention; Behavioral: Volitional intervention; Behavioral: Active Control

INTERVENTIONS:
Behavioral: Motivational intervention — The motivational intervention promotes positive outcome expectancies on physical activity.
Behavioral: Volitional intervention — The volitional intervention promotes the formulation of action plans for physical activity.
Behavioral: Active Control — Participants receive a quiz on physical activity and sports.

SUMMARY:
The purpose of this study is to increase regular physical activity among students by fostering self-management competencies. The intervention was implemented as paper-pencil intervention. The aim of this research project is to evaluate a motivational and volitional intervention in comparison to a control intervention.

Study participants will be recruited in lectures at Freie Universitaet Berlin and followed up twice (two and ten weeks after baseline).

The motivational intervention is expected to increase unmotivated participants' intention to be physically active. The volitional intervention is expected to promote physical activity among motivated but inactive participants. Both interventions are hypothesized to improve self-management competencies over time.

DETAILED DESCRIPTION:
An experimental study is planned over a time period of ten weeks. In the physical activity study, participants will randomly be allocated to either one of two intervention groups (IG) or to an active control group (ACG), receiving a quiz on physical activity and sports. Intervention group 1 receives a paper-pencil intervention which focuses on positive outcome expectancies (motivational intervention). Intervention group 2 receives a paper-pencil intervention which promotes the formulation of action plans for physical activity (volitional intervention).

Furthermore, all participants will receive two emails as intervention boosters until the end of the study.

Study participants will be invited to take part in the study during lectures of the Freie Universitaet Berlin. The students will be followed up twice: two weeks after T1 (paper-pencil), T2 will take place (paper-pencil). Eight weeks after T2 the T3 assessment will be conducted online.

The hypotheses are:

Participants of the motivational intervention report a larger increase in motivation to adopt physical activity from T1 to T2 and T3, as compared to the participants of the volitional or the control intervention. Effects will be larger in unmotivated participants than in already motivated participants.

Participants of the volitional intervention report a larger increase in physical activity from T1 to T2 and T3, as compared to the participants of the motivational or the control intervention. Effects will be larger in motivated participants than in unmotivated participants.

ELIGIBILITY:
Inclusion Criteria:

* to be capable of exercising on their own at a minimum level
* able to fill out a questionnaire (no illiteracy)
* adequate German language ability

Exclusion Criteria:

* no internet access
* no email address

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Self-reported physical activity frequency and duration | two months
  Participants will be asked on how many days per week they were physically active and how much time they had spent on average performing these activities on each of these days (adapted version of the Godin scale)

SECONDARY OUTCOMES:
Algorithm for Stages of Change (SOC) based on behavior and intention | two months
  Participants will be asked if they already are physically active and if they want to be more physically active, using a validated staging algorithm.
Social Cognition | two months
  We will assess social cognition based on a validated psychometric scale that is worded in a behavior-specific manner (physical activity) and has several subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Schwarzer, PhD, Study Chair — Freie Universität Berlin
Locations (1):
- Freie Universität Berlin, Berlin, Germany